CLINICAL TRIAL: NCT03516409
Title: Efficacy of a Synbiotic Product (Probiotics + Prebiotics) in the Prevention of Antibiotics-associated Diarrhoea (AAD) in Infants. A Multicenter, Double Blind, Parallel Group, Placebo Controlled, Randomized Study
Brief Title: Bio-Kult Infantis® in AAD Prevention in Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Probiotics International Ltd. (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAD_BKI_001
Record Dates: First submitted 2018-04-19; First posted 2018-05-04 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Acute Otitis Media
Keywords: probiotics; prebiotics; diarrhoea
MeSH Terms: conditions — Otitis Media; Diarrhea

STUDY DESIGN:
Intervention Model Description: Treatment groups: 6 - 35 months old.
  * Bio-Kult Infantis
  * Placebo (maltodextrine DE19)
Masking Description: A multicenter, double blind, parallel group, placebo controlled, randomized study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bio-Kult Infantis (Active Comparator): 1 sachet once a day mixed with milk, water or food.
  Interventions: Dietary Supplement: Biokult
- Placebo (Placebo Comparator): 1 sachet once a day mixed with milk, water or food.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Biokult — Bio-Kult Infantis® is a multi-strain formula containing a probiotic formulation comprising 7 strains of probiotics, high content of Omega-3, Vitamin D3 and Preplex® (50% FOS and 50% gum acacia).
  Each sachet contains:
  * Minimum 1 billion microorganisms per sachet (1 x 109CFU/g), guaranteed throughout the shelf life
  * DHA + EPA: >1mg per sachet
  * Vitamin D3: 2.5mcg per sachet (50% of Nutrient Reference Value). Bio-Kult Infantis® presents itself in the form of a white powder, packaged in sachets of 1 g each
  Arms: Bio-Kult Infantis
Dietary Supplement: Placebo — IP placebo is manufactured so to contain maltodextrin DE19 and have the same organoleptic properties of the active product (similar to the study product in appearance and taste) but without active ingredient. It contains 100% maltodextrin DE19.
  Moreover, placebo sachets are equal in color, shape and weight (1 g) to IP sachets.
  Arms: Placebo

SUMMARY:
Background: antibiotic-associated diarrhoea (AAD) is defined as an acute inflammation of the intestinal mucosa associated to the administration of antibiotics. Its aetiology seems to be linked to the impact of antibiotics on the normal digestive microbiota. Acute otitis media (AOM) is a common paediatric condition and it is one of the most commonly cited indication for antimicrobial therapy in children (amoxicillin + clavulanic acid).

Treatment modalities for AAD are limited because no established treatment exists for non-Clostridium difficile associated AAD, except for discontinuing antibiotic therapy. Measures to prevent AAD include the use of probiotics. The rationale for the use of probiotics in AAD assumes that, considering the pathogenesis of AAD, AAD is associated with disturbance in the normal intestinal microbiota; administrating specific probiotic strains it is possible to normalize unbalanced indigenous microbiota.

Scientific evidence suggests that prebiotics could be beneficial too. Prebiotics can act in synergy with probiotics, being efficacious in suppressing the growth of pathogenic bacteria that may occur during antibiotic therapy.

Study rationale: the principal side effects of treatment with amoxicillin-clavulanate include diarrhoea, vomiting and allergic reactions. Aim of this study is to evaluate the effectiveness of the administration of a synbiotic product, Bio-Kult Infantis®, in the prevention of AAD during a standard therapy with amoxicillin-clavulanate to treat AOM.

Objective: to evaluate the effectiveness of a synbiotic product in the prevention of Antibiotics-Associated Diarrhoea (AAD) during a concomitant standard therapy with amoxicillin / clavulanic acid, also known as co-amoxiclav, to treat Acute Otitis Media (AOM).

Study design: this is a multicenter, double blind, parallel group, placebo controlled, randomized clinical study. 276 children 6 - 35 months old will be enrolled and then randomized into one of the two study groups (Bio-Kult Infantis® + co-amoxiclav standard treatment for AOM / placebo + co-amoxiclav standard treatment for AOM). A comparison will be performed to evaluate the effectiveness of a synbiotic product in the prevention of AAD during the concomitant standard therapy with co-amoxiclav.

During the study 4 visits will have to be performed at the study centre, and extra visits will be performed in case of AOM relapse after recovery. The study will last for each patient 38 ± 6 days.

ELIGIBILITY:
Inclusion Criteria:

* 1. Parents / legal guardians signed written informed consent to participate in the study.
* 2. Male and female infants aged 6 - 35 months (6 and 35 inclusive).
* 3. Infants eligible to receive co-amoxiclav to treat AOM according to current Italian guidelines, edited by Società Italiana di Pediatria, 2012.
* 4. Outpatients infants (not hospitalized).
* 5. Infants who have received at least 2 doses of pneumococcal conjugate vaccine.
* 6. Infants diagnosed with Acute Otitis Media (AOM) based on the following three criteria:

  1. onset, within the preceding 48 hours, of symptoms that parents or legal guardians rated with a score of at least 3 on the Acute Otitis Media Severity of Symptoms (AOM - SOS);
  2. presence of middle-ear effusion;
  3. moderate or marked bulging of the tympanic membrane or slight bulging accompanied by either otalgia or marked erythema of the membrane
* 7. Infants already exposed to formula milk without Cow Milk Protein Allergy (CMPA) (not requiring a formal diagnosis of CMPA).

Exclusion Criteria:

* 1. Infants with any other acute illness apart from AOM (e.g. pneumonia) or with any other chronic illness (e.g. cystic fibrosis).
* 2. Infants with a clinical history positive for any allergy or intolerance to amoxicillin, clavulanic acid or any component of the active product, the placebo or of the rescue medication (acetaminophen).
* 3. Infants presenting contraindications to the study products, to co-amoxiclav or to the rescue medication, according to concerning Summaries of Product Characteristics (SPC).
* 4. Infants being treated with any drug whose pharmacokinetics can interfere with the intake of amoxicillin, clavulanic acid, the study products or the rescue medication or with any drug with which amoxicillin, clavulanic acid, the study products or the rescue medication can interact, according to concerning Summaries of Product Characteristics (SPC).
* 5. Infants with a clinical history positive for allergy to any other antibiotics.
* 6. Infants who have received antibiotics within 8 weeks prior to enrollment.
* 7. Infants who have had otalgia for longer than 48 hours or perforation of the tympanic membrane.
* 8. Infants suffering from active diarrhoea at time of enrollment or chronic diarrhoea.
* 9. Infants who consumed a probiotic product for medicinal purposes within 7 days prior to enrollment.
* 10. Unwillingness on the part of the parents or legal guardians to interrupt any regular intake of other probiotics during the study period
* 11. Diagnosis of Clostridium difficile-associated diarrhoea (CDAD) within the previous three months from enrolment

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 276 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2018-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of AAD | day 10
  occurrence or non-occurrence of AAD according to time frame. An occurrence of AAD is defined as 3 or more watery stools in 1 day or 2 watery stools daily for at least 2 days

SECONDARY OUTCOMES:
Incidence of AAD | Days 24 and 38
  occurrence or non-occurrence of AAD according to time frame
Duration of AAD | Days 10, 24 and 38
  Frequency (frequency of the occurrences as mean) of AAD according to time frame
Mean stool consistency during antibiotic treatment | from end of antibiotic treatment to Day 2, and from Day 24 to Day 38
  Stool consistency evaluated according to the validated Infatl Stool Scale; mean values will be considered according to time frame
Mean stool frequency | Days 10, 24 and 38
  Frequency of evacuations (frequency of the occurrences per 24 hours)
Incidence and mean frequency of abdominal pain, nausea, vomiting, bloating, and appetite suppression | Days 10, 24 and 38
  Occurrence or non-occurrence and frequency of occurrences as mean according to time frame
Time to resolution of AOM | Day 38
  Time (Days) to the first recording of an Acute Otitis Media Severity of Symptoms score (AOM-SOS Score) of 0 and 1 and the time to the second of two successive recordings of that score according to time frame
Rate of resolution of AOM | Days 10, 24 and 38
  frequency of occurrences (resolution of AOM) as mean according to time frame
Rate of residual middle-ear effusion (fluid behind the tympanic membrane) | Days 10, 24 and 38
  frequency of occurrences (residual middle-ear effusion) as mean according to time frame
Rate of AOM relapse | Days 24 and 38
  frequency of occurrences (AOM relapse) as mean according to time frame
Dermatitis in the diaper area (diaper rash) | Days 10, 24 and 38
  occurrence / or non-occurrence of dermatitis according to time frame
Rate of interruption of antibiotic therapy | Day 10
  occurrence / or non-occurrence according to time frame
Use of acetaminophen (as rescue medication) | Day 38
  Use of acetaminophen according to time frame
Evaluation of product palatability | Day 24
  palatability valuated by parents / legal guardians by means of a VAS according to time frame

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Tripodi, Dr, Principal Investigator — UOC pediatria Hospital "Sandro Pertini"
Locations (1):
- Hospital "Sandro Pertini", Roma, Italia, Italy

IPD SHARING:
Plan to Share IPD: No